CLINICAL TRIAL: NCT05417087
Title: Single Dose Oral Bioequivalence Study of Vortioxetine Hemihydrobromide Orally Disintegrating Tablets 20 mg and 'Trintellix' (Vortioxetine) Tablets 20 mg in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Single Dose Oral Bioequivalence Study of Vortioxetine Hemihydrobromide Orally Disintegrating Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seasons Biotechnology (Taizhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C1B01561
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SF001 administered without water (Experimental): test product administered without water
  Interventions: Drug: Vortioxetine Hemihydrobromide Orally Disintegrating Tablets
- SF001 administered with water (Experimental): test product administered with water
  Interventions: Drug: Vortioxetine Hemihydrobromide Orally Disintegrating Tablets
- Trintellix (Experimental): Reference product administered with water
  Interventions: Drug: Vortioxetine Hydrobromide Tablets

INTERVENTIONS:
Drug: Vortioxetine Hemihydrobromide Orally Disintegrating Tablets — Vortioxetine Hemihydrobromide Orally Disintegrating Tablets 20 mg equivalent to 20 mg of Vortioxetine
  Other Names: SF001 ODT
  Arms: SF001 administered with water; SF001 administered without water
Drug: Vortioxetine Hydrobromide Tablets — Vortioxetine Hydrobromide Tablets 20mg
  Other Names: Trintellix
  Arms: Trintellix

SUMMARY:
An open label, randomized, three-period, three-treatment [Treatment A (test product administered without water), Treatment B (test product administered with water) and Treatment C (Reference product administered with water)], six-sequence, crossover, balanced, single dose oral bioequivalence study.

DETAILED DESCRIPTION:
Single dose oral bioequivalence study of Vortioxetine Hemihydrobromide Orally Disintegrating Tablets 20 mg and 'Trintellix' (Vortioxetine) Tablets 20 mg in healthy adult human subjects under fasting conditions.

* To compare and evaluate the oral bioavailability of Vortioxetine Hemihydrobromide Orally Disintegrating Tablets 20 mg (administered without water and with water) with that of 'Trintellix' (Vortioxetine) Tablets 20 mg in healthy, adult, human subjects under fasting conditions.
* To monitor the safety and tolerability of the subjects.

An open label, randomized, three-period, three-treatment [Treatment A (test product administered without water), Treatment B (test product administered with water) and Treatment C (Reference product administered with water)], six-sequence, crossover, balanced, single dose oral bioequivalence study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25 to 45 years old, both inclusive.
2. Gender: Male and/or non-pregnant, non-lactating female. A. Female of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days prior to first dosing day. They must be using an acceptable form of contraception.

   B. For female of childbearing potential, acceptable forms of contraception include the following:

   i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or ii. Barrier methods containing or used in conjunction with a spermicidal agent, or iii. Surgical sterilization or iv. Practicing sexual abstinence throughout the course of the study.

   C. Female will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

   i. Postmenopausal with spontaneous amenorrhea for at least one year, or ii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or iii. Total hysterectomy and an absence of bleeding for at least 3 months.
3. BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
4. Able to communicate effectively with study personnel.
5. Willing to provide written informed consent to participate in the study.
6. All volunteers must be judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which will include:

   1. A physical examination (clinical examination) with no clinically significant finding.
   2. Results within normal limits or clinically non-significant for the following tests:

      * Additional tests and/or examinations (apart from mentioned in protocol) may be performed, if necessary, based on principal investigator discretion.
      * All results will be assessed against the current laboratory normal ranges at the time of testing and a copy of the normal ranges used will be included in the study documentation.

Exclusion Criteria:

Volunteers must not be enrolled in the study if they meet any one of the following criteria:

1. History of allergic responses to Vortioxetine or other related drugs, or any of its formulation ingredients.
2. Have significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG, chest X-ray recording, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
3. Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
4. History or presence of bronchial asthma.
5. Use of any hormone replacement therapy within 3 months prior to the first dose of study medication.
6. A depot injection or implant of any drug within 3 months prior to the first dose of study medication.
7. Use of CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see http://medicine.iupui.edu/clinpharm/ddis/main-table).
8. History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
9. Smokers who smoke 10 or more cigarettes per day or 20 or more biddies per day or those who cannot refrain from smoking during the study period.
10. History of difficulty with donating blood or difficulty in accessibility of veins.
11. A positive hepatitis screen (includes subtypes B & C).
12. A positive test result for HIV antibody and / or syphilis (RPR).
13. Volunteers who have received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
14. Volunteers who have donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever is greater.
15. History of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.
16. Intolerance to venipuncture
17. Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
18. Institutionalized volunteers.
19. Use of any prescribed medications (including Mono Amine Oxidase Inhibitors, serotonergic antidepressants, nonsteroidal anti-inflammatory drugs (NSAIDs), aspirin, or other drugs that affect coagulation) within 14 days prior to the first dose of study medication.
20. Use of any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
21. Use of grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
22. Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.), cigarettes and tobacco containing products, recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of study medication.
23. Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
24. History of (or have a family history of) bipolar disorder or suicidal thoughts or actions or any other psychiatric problems.
25. History of seizures or convulsions.
26. History of acute narrow-angle glaucoma.
27. Serum sodium value is less than lower limit of normal reference ranges.
28. History of bleeding problems.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Plasma samples will be tested. PK parameter Cmax will be reported. Ratios of PK parameters on SF001 ODT and Trintellix fall within 80.00% to 125.00% | In each period, total 28 blood samples will be collected at pre-dose (0.0 hour) and until 240 hours post dose
  PK parameters will be determined using a non-compartmental analysis. T/R ratio will be reported for Cmax. Ln-transformed Cmax should be within 80.00% to 125.00% with 90% confidence intervals as bioequivelence
Plasma samples will be tested. PK parameter AUCi will be reported. Ratios of PK parameters on SF001 ODT and Trintellix fall within 80.00% to 125.00% | In each period, total 28 blood samples will be collected at pre-dose (0.0 hour) and until 240 hours post dose
  PK parameters will be determined using a non-compartmental analysis. T/R ratio will be reported for AUCi. Ln-transformed AUCi should be within 80.00% to 125.00% with 90% confidence intervals as bioequivelence

CONTACTS AND LOCATIONS:
Overall Officials: Mayur Soni, Ph.D., Principal Investigator — Cliantha Research Limited
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No